CLINICAL TRIAL: NCT06137079
Title: "Iron Overload and Endocrinological Diseases"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Responsible Party: Principal Investigator, Vincenzo Rochira, Professor, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 24/13
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Iron Overload; Thalassemia Major; Thalassemia Intermedia; Hemochromatosis; Endocrinopathy
MeSH Terms: conditions — Iron Overload; beta-Thalassemia; Hemochromatosis; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with hemochromatosis or Thalassemia develop progressive tissue and organs damages secondary to iron overload. Iron overload can result both from transfusional hemosiderosis and excess gastrointestinal iron absorption. Iron deposition in the heart, liver, and multiple endocrine glands results in severe damage to these organs, with variable degrees of endocrine and organ failure.

Although patients with iron overload often present endocrine disorders, the pathogenetic mechanisms underlying endocrinopathies are not completely clear. In particular it is not elucidated if the spectrum of endocrinopathies could change with advancing age. All endocrinological comorbidities can develop from a primary damage of the target gland, from pituitary secondary failure or from both.

The aim of this study is to investigate the prevalence of endocrinological diseases in adult patients with iron overload due to β-thalassemia or hemochromatosis and their impact on well-being and quality of life.

The study design is a prospective cross-sectional clinical study. All subjects enrolled will be evaluated for the endocrine diseases. The study protocol will include data collection from family and patients' history of diseases, physical examination, hormonal assessment for all endocrine axes and instrumental examinations.

The results will provide evidence on the prevalence of endocrine diseases in patients with iron overload and will add information to characterize the type and the degree of endocrine deficiencies, and on the pathogenic mechanisms involved, in order to individualize diagnostic and therapeutic approaches.

ELIGIBILITY:
Inclusion Criteria:

* Certain diagnosis of β-thalassemia major or intermedia
* Certain diagnosis of Hereditary Hemochromatosis
* Adult patients with an age between 18 and 65 years

Exclusion Criteria:

* Subjects with an age < 18 and > 65 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a confirmed diagnosis of β-thalassemia (major or intermedia) or with a diagnosis of hemochromatosis enrolled at the "Unit of Endocrinology, Department of Medical Specialties, Azienda Ospedaliero-Universitaria di Modena Policlinico di Modena, Ospedale Civile di Baggiovara, Modena, Italy".
  Since thalassemia is a rare pathology and considering that the involvement of the endocrine glands in thalassemic patients is extremely common (it is expected to find at least one impaired endocrinological axis in each patient), the number of patients the investigators will enroll is appropriate to make an estimation of the prevalence of endocrine deficiency. Patients will be considered eligible according to the inclusion and exclusion criteria, independently from the presence/absence of known endocrine diseases and after providing their informed signed consent.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2013-06-20; Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Estimate prevalence of endocrine comorbidities of β-thalassemia in adulthood | 12 years

SECONDARY OUTCOMES:
Evaluate prevalence of endocrine diseases to characterize the type and the degree of endocrine deficiencies | 12 years
Evaluate incidence of endocrine diseases to characterize the type and the degree of endocrine deficiencies | 12 years
To investigate the relationships among iron status and endocrine alterations in these group of patients | 12 years
To investigate the relationships among iron status and cardiac disease in these group of patients | 12 years
To investigate the relationships among iron status and liver disease in these group of patients | 12 years

CONTACTS AND LOCATIONS:
Locations (1):
- Unit of Endocrinology of Azienza Ospedaliero-Universitaria di Modena, Modena, Italy